CLINICAL TRIAL: NCT00097435
Title: A Multi-Center, Randomized, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Albuferon (Recombinant Human Albumin-Interferon Alfa Fusion Protein) in Combination With Ribavirin in Interferon Treatment Experienced Subjects With Chronic Hepatitis C
Brief Title: A Study of Albuferon With Ribavirin in Interferon Treatment Experienced Subjects With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinical Protocol ALFR-HC-05
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — albuferon; Ribavirin

INTERVENTIONS:
Drug: Albuferon
Drug: Ribavirin

SUMMARY:
This is a Phase 2, multi-center, randomized, open-label study to evaluate the safety, tolerability, and efficacy of Albuferon in subjects with hepatitis C (HEP C) who failed to respond to previous interferon alfa therapy.

ELIGIBILITY:
Major Inclusion Criteria:

* Have a clinical diagnosis of chronic HEP C established on the basis of detectable viral load, as measured by a serum HCV RNA test during the screening period.
* Have previously failed to respond to treatment with any interferon alfa (IFNa) product
* Have compensated liver disease with the following minimum criteria: white blood cell count > 3,000/mm3, absolute neutrophil count (ANC) > 2,000/mm3, platelets > 125,000/mm3, and hemoglobin (Hb) > 13 g/dL for males or > 12 g/dL for females.

Major Exclusion Criteria:

* Evidence of decompensated cirrhosis or portal hypertension.
* Pregnant or lactating female.
* History of any other medical disease or condition that would make the subject (in the opinion of the investigator) unsuitable for the study.
* A current drug or alcohol addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2004-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The major safety endpoints are the common side effects of IFNa therapy including flu-like symptoms, depression, and hematologic abnormalities.

SECONDARY OUTCOMES:
Sustained virologic response (SVR), defined as undetectable virus at 24 weeks after the end of therapy. The primary efficacy assessment is HCV RNA level.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - Mayo Clinic, Phoenix, Arizona
  - University of Florida CRC, Gainesville, Florida
  - University of Florida at Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Metropolitan Research, Fairfax, Virginia